CLINICAL TRIAL: NCT03735940
Title: DeltaScan for the Assessment of Delirium in the Intensive Care: a Multicenter Stepped Wedge Cluster Randomized Trial (Study 1)
Brief Title: Clinical Evaluation Program of DeltaScan (ICU)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The pandemic caused a rising tide phenomenon on our primary outcomes 1) Delirium detection (increased by visit reduction & masked staff) and 2) Admission duration (increased by reorganizations & quarantines 'impact on being discharged)
Sponsor: UMC Utrecht (Other)
Collaborators: Charite University, Berlin, Germany (Other); KU Leuven (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Prolira (Industry); Factory CRO (Industry); Implementation IQ (Unknown); European Union (Other)
Responsible Party: Principal Investigator, A.J.C. Slooter, Professor of Intensive Care Neuropsychiatry, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: FTI-820555-DeltaScan-study1
Record Dates: First submitted 2018-10-24; First posted 2018-11-08 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Delirium
Keywords: Electroencephalography; Intensive Care; Brain disease; Confusion; Neurobehavioral Manifestations; Nervous System Diseases; Signs and Symptoms; Neurocognitive Disorders; Mental Disorders
MeSH Terms: conditions — Delirium; Brain Diseases; Confusion; Neurobehavioral Manifestations; Nervous System Diseases; Signs and Symptoms; Neurocognitive Disorders; Mental Disorders

STUDY DESIGN:
Intervention Model Description: In this study ICU departments will be randomized with respect to the time they will introduce the DeltaScan following a stepped wedge cluster randomization design. All departments apply 'usual care' in combination with a harmonized delirium treatment protocol during the control phase. After this first time period, each new time period a department switches to the intervention period.
  Due to the first wave of the COVID-19 pandemic the stepped wedge planning was interrupted. Where possible the control period and/or intervention, whichever was affected, will be extended. We marked the first wave of the COVID-19 pandemic from the 15th of March until the 15th of May or longer for a few heavily effected sites with a maximum of 6 months. Data collected during this period will not be used for primary analysis, but may be used for specific sub analyses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control phase (No Intervention): no intervention, i.e. care as usual
- Intervention phase (Experimental): experimental intervention: spot monitoring device, i.e. use of DeltaScan
  Interventions: Other: Spot monitoring device, excl. Sham

INTERVENTIONS:
Other: Spot monitoring device, excl. Sham — o During the control phase the 'care as usual' regarding delirium screening is studied. During the intervention phase the DeltaScan will be studied as screening method for delirium. o During the intervention phase the DeltaScan will be used on the exact same moments, i.e. same time and same amount of measures per day, as the screening methods used in the 'care as usual'.
  Arms: Intervention phase

SUMMARY:
Rationale: Delirium, or acute brain failure, presents as an acute confusional state, and is associated with prolonged hospitalization, an increased risk of dementia, institutionalization and mortality, as well as increased costs. Early detection of delirium would allow for early treatment and improved patient outcomes, but delirium is often not recognized and treatment is therefore delayed or not applied at all. Additionally, current screening tools are subjective, so an alternative, more objective diagnostic tool for early delirium detection is desired. The DeltaScan, a CE-certified device to detect delirium using brief EEG recording, has been recently been found have diagnostic properties that outperform the currently used screening tools.

Objective: To quantify the impact of the use of the DeltaScan on patient outcome (detection rate of delirium and duration of admission) in patients with high risk of delirium compared to the currently used delirium screening tools.

Study design: A prospective multicenter stepped wedge cluster randomized trials in (at least) 4 ICU departments.

Study population: Adult patients admitted to an intensive care unit (ICU) with high risk of delirium.

Intervention: During 12 months, patients presenting at the ICU of participating hospitals with an expected stay > 1 day will be included in the study. First, all hospitals will apply 'usual care' to all patients, i.e. standard delirium screening (e.g. the Confusion Assessment Method (CAM)-ICU) or other currently used tools) in combination with a delirium treatment protocol and subsequent management without application of the DeltaScan for a period of 3 months. Then, during a 6 month period, each 2 months, starting at day 0, randomly allocated hospitals will sequentially start to apply the DeltaScan in all eligible patients (intervention period). During the last 3 months of the study all hospitals will participate in the intervention period.

Main study endpoints:

Primary endpoints: delirium detection rate (i.e. proportion of positive assessments according to the delirium detection tool), and duration of admission at ICU. Secondary endpoints: time interval between admission and the first delirium positive assessment, number of days with at least one positive delirium assessment, delirium incidence, hospital mortality, and direct medical costs of hospitalization.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: During the intervention period EEG recordings using the CE-certified DeltaScan will be made using a strip with EEG electrodes that will be mounted to the head using self-adhesive gel. The EEG recording will be performed two to three times daily and takes 3-4 minutes. During the usual care period the patients will receive the standard delirium screening tool for delirium assessment by a nurse. This assessment will be performed two to three times daily and takes 2-4 minutes depending on the screening tools that is used. Since the DeltaScan has shown to have superior diagnostic performance compared to the DSM5 the burden/risk of misclassification is lower than with the current standard for delirium assessment. Based on the above we consider the burden to participants in this study to be minimal.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the ICU department
* At risk of delirium, defined according to local protocol:

ICU patients: when expected stay is > 1 day

Exclusion Criteria:

* Age younger than 18 years.
* Admitted because of a primary neurological or neurosurgical disease.
* Patients who cannot clinically assessed for delirium, e.g. due to a language barrier or deafness.
* Known pre-existing dementia.
* We decided to add an extra exclusion criteria: Patients infected with SARS-CoV-19 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3630 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Delirium detection rate | From date of admission on the ICU until date of discharge from the ICU or death from any cause, whichever came first, assessed up to 12 months
  The detection rate of delirium will be defined as the proportion of delirium positive assessments during conditions that a patient can be assessed for delirium. A positive delirium assessment in the usual care period will be defined as a positive score on the delirium detection tool that is currently used in the participating department according to the protocol of that department. A positive delirium assessment in the intervention period will be defined as a DeltaScan score of 4 or 5.
Length of admission (days) | From date of admission on the ICU until date of discharge from the ICU or death from any cause, whichever came first, assessed up to 12 months
  The duration of admission will be defined as the cumulative duration of ICU admission. The criteria for discharge will be the same in the usual care period and the intervention period.

SECONDARY OUTCOMES:
The time interval between admission (i.e. ICU admission) and the first delirium positive assessment | From date of admission on the ICU until date of discharge from the ICU or death from any cause, whichever came first, assessed up to 12 months
The number of delirium days | From date of admission on the ICU until date of discharge from the ICU or death from any cause, whichever came first, assessed up to 12 months
  This outcomes is defined as the number of days with at least one positive assessment.
Delirium incidence | From date of admission on the ICU until date of discharge from the ICU or death from any cause, whichever came first, assessed up to 12 months
Hospital mortality | From date of admission on the ICU until date of death from any cause, assessed up to 12 months
Direct medical costs of hospitalization | From date of admission on the ICU until date of discharge from the ICU or death from any cause, whichever came first, assessed up to 12 months
  We aim to collect health care consumption in detail for every included patient. This health care consumption for instance consists of number of hospitalization days, medication, diagnostic procedures. These data will be extracted from the hospital systems. General reference prices (open source, National Tariffs) will be applied to this health care consumption to calculate total costs.
Adherence to new delirium treatment protocol | From date of admission on the ICU until date of discharge from the ICU or death from any cause, whichever came first, assessed up to 12 months
  Steps that are taken (e.g. pharmacological or non-pharmacological treatment, consults of specialist etc.) by the hospital staff after a delirium screener gives a delirium positive score.
Duration of mechanical ventilation | From date of admission on the ICU until date of discharge from the ICU or death from any cause, whichever came first, assessed up to 12 months
Hospital length of stay | From date of admission on the ICU until date of discharge from the hospital or death from any cause, whichever came first, assessed up to 12 months
Incidence of ICU re-admission | From date of admission on the ICU until date of discharge from the hospital or death from any cause, whichever came first, assessed up to 12 months
Number of days alive without delirium and without coma (i.e. RASS -3, -4 or -5) in 28 days | From date of admission on the ICU until date of discharge from the ICU or death from any cause, whichever came first, assessed up to 12 months

OTHER OUTCOMES:
Age | From date of admission on the ICU until date of discharge from the ICU or death from any cause, whichever came first, assessed up to 12 months
Sex | From date of admission on the ICU until date of discharge from the ICU or death from any cause, whichever came first, assessed up to 12 months
Type of admission, defined as acute or elective | From date of admission on the ICU until date of discharge from the ICU or death from any cause, whichever came first, assessed up to 12 months
Admitting discipline, defined as medicine, general surgery, cardiology, or cardiothoracic surgery | From date of admission on the ICU until date of discharge from the ICU or death from any cause, whichever came first, assessed up to 12 months
Reason for not using DeltaScan | From date of admission on the ICU until date of discharge from the ICU or death from any cause, whichever came first, assessed up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Numan T, van den Boogaard M, Kamper AM, Rood PJT, Peelen LM, Slooter AJC; Dutch Delirium Detection Study Group. Delirium detection using relative delta power based on 1-minute single-channel EEG: a multicentre study. Br J Anaesth. 2019 Jan;122(1):60-68. doi: 10.1016/j.bja.2018.08.021. Epub 2018 Oct 2. PMID 30579407
- [Background] van der Kooi AW, Zaal IJ, Klijn FA, Koek HL, Meijer RC, Leijten FS, Slooter AJ. Delirium detection using EEG: what and how to measure. Chest. 2015 Jan;147(1):94-101. doi: 10.1378/chest.13-3050. PMID 25166725